CLINICAL TRIAL: NCT05465772
Title: A Study on COVID-19 Patients With Hypertension and/or Kidney Diseases Admitted to Respiratory ICU , Assiut University Hospitals.
Brief Title: Covid-19 Patients With Hypertension and/or Kidney Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Abdelrhman Kotb Said, Doctor, Assiut University
Other Study IDs: covid-19 patients
Record Dates: First submitted 2022-07-18; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: COVID-19; Hypertension; Kidney Diseases
MeSH Terms: conditions — COVID-19; Hypertension; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. correlation between COVID-19 and Hypertension and/or kidney diseases.
2. Assess Assess the effect of COVID-19 on patients with Hypertension and/or kidney diseases.
3. Assess the effect of hypertension and/or kidney diseases on COVID-19 presentation.
4. Assess the outcome of COVID-19 in patients with hypertension and/or kidney diseases

DETAILED DESCRIPTION:
The pandemic situation with the emergence of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) from China has endangered human lives. Coronavirus disease 2019 (COVID-19) is presented with asymptomatic, mild, or severe pneumonia-like symptoms¹.SARS-CoV-2 has infected humans in all age groups, of all ethnicities, both males and females while spreading through communities at an alarming rate². COVID-19 patients with hypertension, chronic kidney disease, Diabetes, malignancies, HIV, and other comorbidities could develop a life-threatening situation. From the data have reported the characteristics of comorbidities in patients with COVID-19, hypertension was present in nearly 21%, followed by diabetes in nearly 11%, and established cardiovascular disease (CVD) in approximately 7% of patients³.

Hypertension posed an increased risk of severe morbidity (approx. 4-fold) and death (approx. 7-fold) from COVID-19 in the presence of multiple comorbidities⁴.

The patients with underlying kidney problems are vulnerable to developing COVID-19 infection.The disease also has had consequences on longitudinal management of patients with chronic kidney disease and end stage kidney disease.

ELIGIBILITY:
Inclusion Criteria:

Patients above 18 years old. Patients who diagnosed as COVID-19 PCR positive with hypertension and/or kidney diseases.

Exclusion Criteria:

Young patients below 18 years old. Patients who refused to participate in reseach

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted to ICU with positive PCR with Hypertension and/or kidney diseases.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Covid-19 and Hypertension and/or kidney diseases | Baseline
  Effect of COVID-19 on patients with Hypertension and/or kidney diseases and assess the outcome of COVID-19 in patients with hypertension and/or kidney diseases.